CLINICAL TRIAL: NCT02737735
Title: The Effect on Decreasing Chemotherapeutic Toxicity and Increasing Anti-tumor Effect of Chinese Herbs Based on Syndrome Differentiation
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Sun Bao-guo, Principal Investigator, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SBao-guo
Record Dates: First submitted 2016-03-26; First posted 2016-04-14 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-03

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemotherapy combined with compound herbal medicine (Experimental): Standard chemotherapy protocols on phase IIIB/IV non-small-cell lung cancer for 24 weeks combined with compound Chinese herbal medicine for 2 years，which include 15 kinds of Chinese herbs:Thunberg fritillary bulb,antimutangenic ,cimicifuga foetida,astragalus,pinellia ,Radix Ophiopogonis ,Solanum nigrum,Hedyotis diffusa,Prunella vulgaris ,cordate houttuynia,Herba Patriniae,dried orange peel ,Codonopsis,Wolfiporia extensa,Coix seed,Rhizoma Alismatis.
  Interventions: Drug: standard chemotherapy medicine combined with Chinese herbs
- Chemotherapy (Active Comparator): The therapy of standard chemotherapy protocols on phase IIIB/IV non-small-cell lung cancer for 24 weeks
  Interventions: Drug: standard chemotherapy medicine

INTERVENTIONS:
Drug: standard chemotherapy medicine combined with Chinese herbs
  Arms: Chemotherapy combined with compound herbal medicine
Drug: standard chemotherapy medicine
  Arms: Chemotherapy

SUMMARY:
To study the effect on decreasing chemotherapeutic toxicity and increasing anti-tumor treatment of Chinese Herbs based on syndrome differentiation

ELIGIBILITY:
Inclusion Criteria:

* Histology and cytology diagnosed IIIB or IV non-small-cell lung cancer (NSCLC) and untreated; Age > 18 ages
* Sex unlimited; ECOG (Eastern Cooperative Oncology Group) fitness score (Performance status, PS)≤2.
* White blood cell count ≥ 3 x 10E9 / L, neutrophils ≥1 x 109 p/L, hemoglobin≥80 g/L , platelet ≥100 x 10E9 / L
* ALT, AST, normal or less than 2 times, bilirubin is normal
* Serum level in the normal range;Thr ecg is normal
* Expected survival time≥ 3 months or more;
* Agreed to the treatment combined traditional Chinese medicine with western medicine

Exclusion Criteria:

* Engaged in other clinical subjects
* Pregnant or lactating women, women in childbearing age refuse contraceptives during the trail
* Severe pneumonia, tuberculosis, lung abscess, myocarditis and other malignant tumor
* Severe damage of heart, liver and kidney (cardiac function grade 3 ~ 4, ALT and/or AST 2 times more than normal , Cr more the normal limit)
* Mental illness, Refused to partner; Cannot obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-03; Primary Completion 2019-12 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival rate | 36months
progression-free survival rate | 36months

OTHER OUTCOMES:
Quality of Life Questionnaire (EORTC QLQ C30)scores | 36months
RECIST(Response Evaluation Criteria In Solid Tumors) | 36months
KPS scores | 36months
nutritional evaluation scores | 36months
BMS(Bone marrow suppression) scores | 36months
Gastrointestinal reactions scores | 36months
hair loss level scores | 36months
AST value | 36months
ALT value | 36months
creatinine value | 36months

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Sun-yat Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No